CLINICAL TRIAL: NCT03158636
Title: Profiling of Oncology Patients as Part of Clinical Care and Research
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Cancer Trials New Zealand, Professor of Oncology, University of Auckland, New Zealand
Other Study IDs: CTNZ-2016-01
Record Dates: First submitted 2017-05-03; First posted 2017-05-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Retrospective tissue collection. Circulating tumour DNA. Prospective tumour biopsies (where feasible).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The era of precision medicine is an exciting time for clinicians, scientists and patients alike. The increasing appreciation and identification of specific mutations that drive cancers, leaves us on the threshold of a new era in which biomarkers will be used to direct targeted agents to only those patients most likely to respond. The potential medical and scientific benefits of such a personalised approach to cancer therapy are immense. However, a number of barriers challenge successful implementation of this approach of which spatial and temporal heterogeneity are a major concern.

Gynaecological cancers are a major cause of mortality and morbidity internationally. In Auckland 150 new patients with ovarian, endometrial or cervical cancer are seen by a medical oncologist each year. In general, when these diseases recur, there are few effective therapeutic options and prognosis is poor. Better therapeutic targets and treatments are an unmet need across these tumour types with treatment paradigms still based upon platinum based therapy.

PROSPER (Profiling of Oncology Patients as part of Clinical care and Research) will investigate the evolution of gynaecological cancers over time and in response to treatment to develop better biomarkers to guide treatment decisions and ultimately improve patient outcomes. Biopsies at relapse will be collected and profiled with a 580 cancer gene panel. Circulating tumour DNA will be collected and analysed alongside biopsies as a potential non-invasive alternative. Linking genomic and clinical data will allow us to learn more to begin to change our paradigm of care.

DETAILED DESCRIPTION:
PROSPER is a pilot project that will assess the ability to integrate genomic results into patient care and research.

All patients will be consented to be involved. Involvement will be completely voluntary. Patients with gynaecological cancers or patients potentially eligible for a phase I trial who are receiving cancer care under medical oncology at Auckland City Hospital will be approached to consider participation in this study. All patients who are over 18 and potentially eligible for further therapy (standard of care or as part of a clinical trial) will be considered.

Patients who agree to participate in PROSPER will provide archived tumour specimens (primary tumour and/or metastasis; tumour block or 15-20 unstained paraffin-embedded slides [minimum of 15 unstained slides if block not available], plus one H&E stained slide). Molecular profiling will be performed at the University of Auckland taking advantage of local expertise. A hybridisation capture DNA sequencing approach obtaining 500x-1000x coverage of a panel of 578 cancer genes will be used. This approach has recently been used to successfully analyse over 40 paired tumour and normal FFPE tissues by Prof. Cristin Print's University of Auckland laboratory (NimbleGen comprehensive cancer panel). Tumour tissue that remains after molecular profiling will be banked (with patients' consent) and may be subject to additional genomic sequencing analysis (e.g. whole genome sequencing), RNA expression analysis (Affymetrix Primeview), protein expression analysis (e.g. Western blot, IHC), and/or DNA copy number analysis (e.g. array CGH, quantitative PCR, FISH) based on resources available. Only validated results of these analyses will be conveyed to treating physicians and made available in patients' records.

Patients must agree to provide whole blood for biobanking. This will provide a source of normal DNA for differentiation of constitutional versus somatic (tumour) molecular changes. Blood samples will also be used to detect circulating tumour DNA to assess this as an alternative to fresh biopsies.

On documentation of relapse patients will be asked (where feasible) to provide a tumour biopsy and blood sample for further profiling. As biopsies become an increasingly common requirement in clinical trials, willingness of patients, procedural safety and useful tissue acquisition are critical elements of success. In patients with high grade serous ovarian cancer research biopsies have been shown to be safe, and feasible. In this project, investigators will collect ctDNA (circulating tumour DNA) alongside tumour biopsies to allow correlation and validation of the role of ctDNA as a non-invasive alternative to biopsies. Relating baseline expression profiles to treatment outcomes for each patient will help optimise drug therapy by improving patient selection and monitoring. This project will build upon plasma genomic initiatives already underway in breast, colorectal, and neuroendocrine cancers.

All decision making about the advisability of biopsy and site to be sampled will be at the discretion of the clinician(s) who have primary care responsibility for the participants. The possible risks and benefits of obtaining additional fresh tumour samples at the time of relapse or emergence of drug resistance, will be fully explained to the patient. Consent to undergo a biopsy to obtain fresh tumour will be entirely voluntary and will not affect the patient's eligibility to participate in PROSPER or to participate in a related clinical trial. Participants will be allowed to decline biopsies at any stage, even if they have consented previously. Biopsies at relapse may be taken surgically or radiologically depending on feasibility and what other interventions are being undertaken as part of standard of care. A small proportion of these patients with isolated relapse may undergo surgery and in this scenario samples will be collected at this time. If biopsies are to be done radiologically, at least three 14-16 gauge core tumour biopsies will be collected.

PROSPER will assess the clinical significance and feasibility of a profiling programme. Measures of benefit will include the percentage of patients treated as part of a clinical trial; number of patients receiving targeted therapy based on molecular aberrations; and integration of molecular information in practice. The study aims to profile 50-100 patients in the first year. In Auckland Hospital, 150 new patients with ovarian, cervical or endometrial cancer are treated annually. Additionally, 100-150 patients with relapsed disease are treated each year. This creates a large population that will be eligible for this project.

A secure PROSPER database to register patients' clinical details will be established. Throughout the study's duration, data management processes will be followed in accordance with local SOPs, in an effort to maximise data quality and security.

The registry will be password protected and accessible to registered users only. Doctors referring patients for enrolment in PROSPER will be able to view each of their patient's results in an identifiable format for use in clinical decision making. Other registered doctors will be able to see all other patient details in a de-identified manner allowing them to view clinical details and assay results of like patients. If patients' information is sent overseas as part of the study, only de-identified data will be sent.

Appropriate steps will be taken to protect health information against loss, unauthorised access, use, modification, or disclosure or other misuse. For collection of tissue, patient information will be de-identified and a new unique alpha-numeric identifier will be assigned to each participant for all tissue specimens. Identification of individuals will be possible only by reference to a master index, which will be kept on hard copy in a locked file in a secure area, and on a password-protected encrypted database. If tissue or isolated molecular products are sent overseas for specialised scientific studies, only the anonymised study ID would be provided.

Clinical data will be collected by the principal investigator, project manager, local clinical lead or other health professional under the approval of the local clinical lead, from patients' medical records into a password protected central database housed on a secure server under responsibility of the University of Auckland. All data will be de-identified at the point of extraction from the database prior to any analysis.

No directly identifiable information will be included in publications arising from this study, nor will NHI numbers, dates of birth, or names of donors be shared with collaborators, with the exception of collaborators involved in the care of the patient.

Clinicians involved with patient care will have access to the profiling results if patients have provided consent for this.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histological diagnosis of gynaecological cancer OR diagnosis of cancer and candidate for phase I clinical trial
3. ECOG performance status ≤2
4. Life expectancy of greater than 3 month
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Any contraindication to biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gynaecological cancers or those patients potentially eligible for a phase I trial who are receiving cancer care under medical oncology at Auckland City Hospital will be approached to consider participation in this study. All patients who are over 18 and potentially eligible for further therapy (standard of care or as part of a clinical trial) will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Utilisation rates of molecular profiling information. | 3 years

SECONDARY OUTCOMES:
Number of patients where the molecular profiling information guided standard treatment or clinical trial enrollment. | 3 years
Clinical trial accrual rates among patients with available molecular profiling data. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Wilson, MBChb, FRACP, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- University of Auckland / Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be available for other research through applications to the governance committee of PROSPER. Applications will require ethics approval.
Supporting Information: Study Protocol
Time Frame: to be confirmed
Access Criteria: Deidentified patient data will be available for other research through applications to the governance committee of PROSPER. Applications will require ethics approval.